CLINICAL TRIAL: NCT00443703
Title: A Multicenter, Double-Blind, Randomized, Active-Controlled Study to Evaluate the Safety and Antiretroviral Activity of MK0518 Versus KALETRA in HIV-Infected Patients Switched From a Stable KALETRA-Based Regimen - Study A
Brief Title: MK0518 in the Treatment of HIV-Infected Patients Switched From a Protease Inhibitor Regimen (0518-032)(TERMINATED)
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: primary efficacy analysis at Week 24 did not demonstrate non-inferiority of raltegravir versus lopinavir (+) ritonavir
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0518-032; 2007_507
Record Dates: First submitted 2007-03-02; First posted 2007-03-06 (Estimated); Results first posted 2009-12-01 (Estimated); Last update posted 2017-03-21 (Actual); Status verified 2017-02

CONDITIONS: HIV Infection
Keywords: treatment experienced
MeSH Terms: conditions — HIV Infections | interventions — Raltegravir Potassium; Lopinavir; Ritonavir; lopinavir-ritonavir drug combination

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- 1 (Experimental): Arm 1: MK0518 (raltegravir) + placebo to KALETRA™ (lopinavir (+) ritonavir )
  Interventions: Drug: MK0518 (raltegravir); Drug: Comparator: placebo
- 2 (Active Comparator): Arm 2: KALETRA™ (lopinavir (+) ritonavir) + placebo to MK0518 (raltegravir)
  Interventions: Drug: Comparator: KALETRA™ (lopinavir (+) ritonavir ); Drug: Comparator: placebo

INTERVENTIONS:
Drug: MK0518 (raltegravir) — MK0518 (raltegravir) 400 mg by mouth (PO) twice daily (b.i.d) for up to 48 weeks of treatment
  Other Names: MK0518; raltegravir
  Arms: 1
Drug: Comparator: KALETRA™ (lopinavir (+) ritonavir ) — KALETRA™ (lopinavir (+) ritonavir ) 400/100 mg by mouth (PO) twice daily (b.i.d.) for up to 48 weeks of treatment.
  Other Names: KALETRA
  Arms: 2
Drug: Comparator: placebo — MK0518 (raltegravir) 400 mg by mouth (PO) twice daily (b.i.d.) Placebo for up to 48 weeks of treatment
  Arms: 2
Drug: Comparator: placebo — KALETRA™ (lopinavir (+) ritonavir ) 400/100 mg by mouth (PO) twice daily (b.i.d.) Placebo for up to 48 weeks of treatment.
  Arms: 1

SUMMARY:
The purpose of this study is to investigate the efficacy, safety, and tolerability of an investigational treatment for patients with HIV.

ELIGIBILITY:
Inclusion Criteria:

* Patient is at least 18 years of age
* Patient is Human Immunodeficiency Virus (HIV) positive
* Patient has documented Human Immunodeficiency Virus (HIV) RiboNucleic Acid (RNA) <50 copies/milliliter (mL) for at least 3 months while on a KALETRA based regimen
* Patient has been on a KALETRA based regimen for at least 3 months without a change in background antiretroviral therapy
* Patient has no documentation of HIV RNA >50 copies/mL for at least 3 months while on the KALETRA based regimen

Exclusion Criteria:

* Patient is or plans to become pregnant, or nursing a child
* Patient plans to donate eggs or impregnate/donate sperm
* Patient is receiving Stavudine (d4T) as a component of the background antiretroviral therapy
* Patient is currently receiving a second protease inhibitor in addition to KALETRA
* Patient is currently receiving, or has received in the past twelve weeks, treatment for the management of elevated lipids
* Patient has used another experimental HIV-integrase inhibitor
* Patient has a current (active) diagnosis of acute hepatitis due to any cause
* Patient has used systemic immunosuppressive therapy within one month prior to treatment in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 352 (Actual)
Dates: Start 2007-05; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
http://www.merck.com/clinical-trials/pdf/Merck%20Procedure%20on%20Clinical%20Trial%20Data%20Access%20Final_Updated%20July_9_2014.pdf
  http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Derived] Eron JJ, Young B, Cooper DA, Youle M, Dejesus E, Andrade-Villanueva J, Workman C, Zajdenverg R, Fatkenheuer G, Berger DS, Kumar PN, Rodgers AJ, Shaughnessy MA, Walker ML, Barnard RJ, Miller MD, Dinubile MJ, Nguyen BY, Leavitt R, Xu X, Sklar P; SWITCHMRK 1 and 2 investigators. Switch to a raltegravir-based regimen versus continuation of a lopinavir-ritonavir-based regimen in stable HIV-infected patients with suppressed viraemia (SWITCHMRK 1 and 2): two multicentre, double-blind, randomised controlled trials. Lancet. 2010 Jan 30;375(9712):396-407. doi: 10.1016/S0140-6736(09)62041-9. Epub 2010 Jan 12. PMID 20074791

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Phase III; First Patient In: 20-Jun-2007; Last Patient Last Visit for Week 24 (primary endpoint): 31-Oct-2008
  47 Sites (US, Canada, Denmark, Germany, Italy, Portugal, Spain, United Kingdom, and Australia).
Pre-assignment Details: HIV-seropositive patients who were ≥18 years old, had documented HIV RNA <50 copies/mL for at least 3 months, had been on a KALETRA™-based regimen for at least 3 months without a change in background antiretroviral therapy, and had no documentation of HIV RNA >50 copies/mL for at least 3 months.
Groups:
- MK0518 400 mg b.i.d.: MK0518 400 mg, which can be taken by mouth (PO) twice a day (b.i.d.), approximately 12 hours (10 to 14 hours) apart without regard to food, and placebo to KALETRA™ , which can be taken by mouth (PO) twice a day (b.i.d.), approximately 12 hours (10 to 14 hours) apart without regard to food
- KALETRA™ 400/100 mg b.i.d.: KALETRA™ 400/100 mg, which can be taken by mouth (PO) twice a day (b.i.d.), approximately 12 hours (10 to 14 hours) apart without regard to food, and placebo to MK0518 , which can be taken by mouth (PO) twice a day (b.i.d.), approximately 12 hours (10 to 14 hours) apart without regard to food
Period: Overall Study
Arm/Group | MK0518 400 mg b.i.d. | KALETRA™ 400/100 mg b.i.d.
Started | 177 | 175
Treated | 174 | 174
Completed | 149 | 157
Not Completed | 28 | 18
Not completed — Never Treated | 3 | 1
Not completed — Adverse Event | 7 | 3
Not completed — Lack of Efficacy | 3 | 1
Not completed — Lost to Follow-up | 0 | 4
Not completed — Physician Decision | 4 | 2
Not completed — Protocol Violation | 1 | 1
Not completed — Withdrawal by Subject | 9 | 6
Not completed — Progressive Disease | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MK0518 400 mg b.i.d. | KALETRA™ 400/100 mg b.i.d. | Total
Number analyzed (Participants) | 174 | 174 | 348
Age, Continuous [Mean (Full Range); unit: years] | 44.4 [23 to 70] | 43.6 [24 to 71] | 44.0 [23 to 71]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 45 | 73
  Male | 146 | 129 | 275
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 25 | 23 | 48
  Not Hispanic or Latino | 149 | 151 | 300
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 3 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 24 | 28 | 52
  White | 146 | 141 | 287
  More than one race | 2 | 2 | 4
  Unknown or Not Reported | 0 | 0 | 0
Cluster of Differentiation 4 (CD4) Cell Count [Mean (Full Range); unit: cells/mm3] | 477.6 [65 to 1446] | 508.2 [87 to 1510] | 492.9 [65 to 1510]
Fasting (non-random) serum High Density Lipoprotein-Cholesterol (HDL-C) [Mean (Standard Deviation); unit: mg/dL] | 48.8 (16.4) | 47.1 (14.0) | 47.9 (15.2)
Fasting (non-random) serum Low Density Lipoprotein-Cholesterol (LDL-C) [Mean (Standard Deviation); unit: mg/dL] | 115.3 (40.3) | 104.8 (35.9) | 110.0 (38.5)
Fasting (non-random) serum cholesterol [Mean (Standard Deviation); unit: mg/dL] | 215.3 (48.2) | 203.9 (52.3) | 209.6 (50.6)
Fasting (non-random) serum triglyceride [Mean (Standard Deviation); unit: mg/dL] — Standard Deviation (Robust): calculated as interquartile range (IQR)/1.075, where IQR=3rd quartile-1st quartile.
  mg/dL | 189.5 (134.0) | 162.0 (112.6) | 175.0 (126.5)
Non-HDL-C [Mean (Standard Deviation); unit: mg/dL] | 165.5 (48.5) | 156.8 (53.0) | 161.1 (50.9)

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Plasma Human Immunodeficiency Virus (HIV) RiboNucleic Acid (RNA) <50 Copies/mL at Week 24
Time Frame: Week 24
Population: Full analysis set; two patients were excluded from the analysis because they did not have an HIV RNA test performed at Week 24 but had a test result of HIV RNA <50 copies/mL at Week 12 and Week 36.
Measure: Number; unit: Participants
Arm/Group | MK0518 400 mg b.i.d. | KALETRA™ 400/100 mg b.i.d.
Number analyzed (Participants) | 172 | 174
Participants | 139 | 152

2. Primary Outcome: Number of Patients With Clinical Adverse Experiences (CAEs) Through 24 Weeks
Description: An adverse experience is defined as any unfavorable and unintended change in the structure, function, or chemistry of the body temporally associated with the use of the SPONSOR'S (Merck & Co., Inc.) product, whether or not considered related to the use of the product
Time Frame: 24 Week last patient last visit
Population: All patients who took study medication were included in the analysis
Measure: Number; unit: Participants
Arm/Group | MK0518 400 mg b.i.d. | KALETRA™ 400/100 mg b.i.d.
Number analyzed (Participants) | 174 | 174
Participants
  With CAEs | 109 | 106
  Without CAEs | 65 | 68

3. Other Pre Specified Outcome: Number of Patients With Serious CAEs Through 24 Weeks
Description: Serious CAEs are any AEs occurring at any dose that; results in death; or is life threatening; or results in a persistent or significant disability/incapacity; or results in or prolongs an existing inpatient hospitalization; or is a congenital anomaly/birth defect; or is a cancer; or is an overdose
Time Frame: 24 Week last patient last visit
Population: All patients who took study medication were included in the analysis
Measure: Number; unit: participants
Arm/Group | MK0518 400 mg b.i.d. | KALETRA™ 400/100 mg b.i.d.
Number analyzed (Participants) | 174 | 174
participants
  With Serious CAEs | 15 | 10
  Without Serious CAEs | 159 | 164

4. Other Pre Specified Outcome: Number of Patients With Drug-related CAEs Through 24 Weeks
Description: Patients with drug-related (as assessed by an investigator who is a qualified physician, according to his/her best clinical judgement) CAEs.
Time Frame: 24 Week last patient last visit
Population: All patients who took study medication were included in the analysis
Measure: Number; unit: participants
Arm/Group | MK0518 400 mg b.i.d. | KALETRA™ 400/100 mg b.i.d.
Number analyzed (Participants) | 174 | 174
participants
  With drug-related CAEs | 24 | 19
  Without drug-related CAEs | 150 | 155

5. Other Pre Specified Outcome: Number of Patients With Serious Drug-related CAEs Through 24 Weeks
Description: Serious CAEs are any AEs occurring at any dose that; results in death; or is life threatening; or results in a persistent or significant disability/incapacity; or results in or prolongs an existing inpatient hospitalization; or is a congenital anomaly/birth defect; or is a cancer; or is an overdose. Drug-related are as assessed by an investigator who is a qualified physician, according to his/her best clinical judgement
Time Frame: 24 Week last patient last visit
Population: All patients who took study medication were included in the analysis
Measure: Number; unit: participants
Arm/Group | MK0518 400 mg b.i.d. | KALETRA™ 400/100 mg b.i.d.
Number analyzed (Participants) | 174 | 174
participants
  With Serious drug-related CAEs | 0 | 0
  Without Serious drug-related CAEs | 174 | 174

6. Other Pre Specified Outcome: Number of Patients That Died by 24 Week Last Patient Last Visit
Time Frame: 24 Week last patient last visit
Population: All patients who took study medication were included in the analysis
Measure: Number; unit: participants
Arm/Group | MK0518 400 mg b.i.d. | KALETRA™ 400/100 mg b.i.d.
Number analyzed (Participants) | 174 | 174
participants
  Died | 0 | 0
  Did Not Die | 174 | 174

7. Other Pre Specified Outcome: Number of Patients That Discontinued Due to CAEs Through 24 Weeks
Time Frame: 24 Week last patient last visit
Population: All patients who took study medication were included in the analysis
Measure: Number; unit: participants
Arm/Group | MK0518 400 mg b.i.d. | KALETRA™ 400/100 mg b.i.d.
Number analyzed (Participants) | 174 | 174
participants
  Discontinued with CAEs | 4 | 4
  Did not Discontinue with CAEs | 170 | 170

8. Other Pre Specified Outcome: Number of Patients That Discontinued Due to Drug Related CAEs Through 24 Weeks
Time Frame: 24 Week last patient last visit
Population: All patients who took study medication were included in the analysis
Measure: Number; unit: participants
Arm/Group | MK0518 400 mg b.i.d. | KALETRA™ 400/100 mg b.i.d.
Number analyzed (Participants) | 174 | 174
participants
  Discontinued with drug related CAEs | 2 | 3
  Did Not Discontinue with drug related CAEs | 172 | 171

9. Other Pre Specified Outcome: Number of Patients With Laboratory Adverse Experiences (LAEs) Through 24 Weeks
Description: A laboratory adverse experience (LAE) is defined as any unfavorable and unintended change in the chemistry of the body temporally associated with the use of the SPONSOR'S (Merck & Co., Inc.) product, whether or not considered related to the use of the product
Time Frame: 24 Week last patient last visit
Population: All patients who took study medication were included in the analysis
Measure: Number; unit: participants
Arm/Group | MK0518 400 mg b.i.d. | KALETRA™ 400/100 mg b.i.d.
Number analyzed (Participants) | 174 | 174
participants
  With LAEs | 11 | 7
  Without LAEs | 163 | 167

10. Other Pre Specified Outcome: Number of Patients With Drug-related Laboratory Adverse Experiences (LAEs) Through 24 Weeks
Description: Patients with drug-related (as assessed by an investigator who is a qualified physician, according to his/her best clinical judgement) LAEs
Time Frame: 24 Week last patient last visit
Population: All patients who took study medication were included in the analysis
Measure: Number; unit: participants
Arm/Group | MK0518 400 mg b.i.d. | KALETRA™ 400/100 mg b.i.d.
Number analyzed (Participants) | 174 | 174
participants
  With LAEs | 6 | 2
  Without LAEs | 168 | 172

11. Other Pre Specified Outcome: Number of Patients With Serious LAEs Through 24 Weeks
Description: Serious LAEs are any LAEs occurring at any dose that; results in death; or is life threatening; or results in a persistent or significant disability/incapacity; or results in or prolongs an existing inpatient hospitalization; or is a congenital anomaly/birth defect; or is a cancer; or is an overdose
Time Frame: 24 Week last patient last visit
Population: All patients who took study medication were included in the analysis
Measure: Number; unit: participants
Arm/Group | MK0518 400 mg b.i.d. | KALETRA™ 400/100 mg b.i.d.
Number analyzed (Participants) | 174 | 174
participants
  With LAEs | 0 | 0
  Without LAEs | 174 | 174

12. Other Pre Specified Outcome: Number of Patients That Discontinued Due to LAEs Through 24 Weeks
Time Frame: 24 Week last patient last visit
Population: All patients who took study medication were included in the analysis
Measure: Number; unit: participants
Arm/Group | MK0518 400 mg b.i.d. | KALETRA™ 400/100 mg b.i.d.
Number analyzed (Participants) | 174 | 174
participants
  Discontinued with LAEs | 2 | 1
  Did Not Discontinue with LAEs | 172 | 173

13. Other Pre Specified Outcome: Number of Patients That Discontinued With Drug Related LAEs Through 24 Weeks
Description: Number of patients that discontinued with drug-related (as assessed by an investigator who is a qualified physician, according to his or her clinical judgement) LAEs.
Time Frame: 24 Week last patient last visit
Population: All patients who took study medication were included in the analysis
Measure: Number; unit: participants
Arm/Group | MK0518 400 mg b.i.d. | KALETRA™ 400/100 mg b.i.d.
Number analyzed (Participants) | 174 | 174
participants
  Discontinued with Drug Related LAEs | 2 | 1
  Did Not Discontinue with Drug Related LAEs | 172 | 173

14. Primary Outcome: Mean Percent Change From Baseline in Fasting Serum Cholesterol at Week 12
Time Frame: Baseline and Week 12
Population: Patients who had both baseline and at least one post-baseline measurement were included in the analysis
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | MK0518 400 mg b.i.d. | KALETRA™ 400/100 mg b.i.d.
Number analyzed (Participants) | 142 | 146
Percent Change | -12.83 (12.19) | 0.70 (14.69)

15. Primary Outcome: Mean Percent Change From Baseline in Non-High-Density Lipoprotein Cholesterol (Non-HDL-C) at Week 12
Time Frame: Baseline and Week 12
Population: Patients who had both baseline and at least one post-baseline measurement were included in the analysis
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | MK0518 400 mg b.i.d. | KALETRA™ 400/100 mg b.i.d.
Number analyzed (Participants) | 140 | 145
Percent Change | -15.17 (15.80) | 2.31 (19.37)

16. Primary Outcome: Mean Percent Change From Baseline in Fasting Serum Low-Density Lipoprotein Cholesterol (LDL-C) at Week 12
Time Frame: Baseline and Week 12
Population: Patients who had both baseline and at least one post-baseline measurement were included in the analysis
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | MK0518 400 mg b.i.d. | KALETRA™ 400/100 mg b.i.d.
Number analyzed (Participants) | 134 | 135
Percent Change | -2.43 (22.63) | 2.05 (29.87)

17. Primary Outcome: Mean Percent Change From Baseline in Fasting Serum High-Density Lipoprotein Cholesterol (HDL-C) at Week 12
Time Frame: Baseline and Week 12
Population: Patients who had both baseline and at least one post-baseline measurement were included in the analysis
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | MK0518 400 mg b.i.d. | KALETRA™ 400/100 mg b.i.d.
Number analyzed (Participants) | 140 | 145
Percent Change | -0.86 (18.71) | 0.78 (25.38)

18. Primary Outcome: Median Percent Change From Baseline in Serum Triglyceride at Week 12
Description: Standard Deviation (Robust): calculated as interquartile range (IQR)/1.075, where IQR=3rd quartile-1st quartile.
Time Frame: Baseline and Week 12
Population: Patients who had both baseline and at least one post-baseline measurement were included in the analysis
Measure: Median (Standard Deviation); unit: Percent Change
Arm/Group | MK0518 400 mg b.i.d. | KALETRA™ 400/100 mg b.i.d.
Number analyzed (Participants) | 142 | 146
Percent Change | -41.50 (35.37) | 3.56 (59.36)

19. Secondary Outcome: Mean Percent Change From Baseline in Fasting Serum Cholesterol at Week 24
Time Frame: Baseline and Week 24
Population: Patients who had both baseline and at least one post-baseline measurement were included in the analysis
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | MK0518 400 mg b.i.d. | KALETRA™ 400/100 mg b.i.d.
Number analyzed (Participants) | 146 | 149
Percent Change | -13.81 (12.02) | 2.70 (17.69)

20. Secondary Outcome: Mean Percent Change From Baseline in Non-High-Density Lipoprotein Cholesterol (Non-HDL-C) at Week 24
Time Frame: Baseline and Week 24
Population: Patients who had both baseline and at least one post-baseline measurement were included in the analysis
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | MK0518 400 mg b.i.d. | KALETRA™ 400/100 mg b.i.d.
Number analyzed (Participants) | 143 | 148
Percent Change | -15.03 (16.52) | 5.53 (21.96)

21. Secondary Outcome: Mean Percent Change From Baseline in Fasting Serum Low-Density Lipoprotein Cholesterol (LDL-C) at Week 24
Time Frame: Baseline and Week 24
Population: Patients who had both baseline and at least one post-baseline measurement were included in the analysis
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | MK0518 400 mg b.i.d. | KALETRA™ 400/100 mg b.i.d.
Number analyzed (Participants) | 139 | 143
Percent Change | -1.12 (23.66) | 8.54 (27.44)

22. Secondary Outcome: Mean Percent Change From Baseline in Fasting Serum High-Density Lipoprotein Cholesterol (HDL-C) at Week 24
Time Frame: Baseline and Week 24
Population: Patients who had both baseline and at least one post-baseline measurement were included in the analysis
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | MK0518 400 mg b.i.d. | KALETRA™ 400/100 mg b.i.d.
Number analyzed (Participants) | 143 | 148
Percent Change | -4.42 (17.80) | -1.70 (20.24)

23. Secondary Outcome: Median Percent Change From Baseline in Serum Triglyceride at Week 24
Description: Standard Deviation (Robust): calculated as interquartile range (IQR)/1.075, where IQR=3rd quartile-1st quartile.
Time Frame: Baseline and Week 24
Population: Patients who had both baseline and at least one post-baseline measurement were included in the analysis
Measure: Median (Standard Deviation); unit: Percent Change
Arm/Group | MK0518 400 mg b.i.d. | KALETRA™ 400/100 mg b.i.d.
Number analyzed (Participants) | 146 | 149
Percent Change | -44.53 (31.43) | 6.14 (57.80)

ADVERSE EVENTS:
Time Frame: Adverse experiences that occurred after randomization and through Week 24 last patient last visit (31-Oct-2008) were collected.
Description: The list of Other Adverse Events has an incidence cut off of 2%, includes clinical as well laboratory Adverse Events, and does not include Serious Adverse Events.
Arm/Group | MK0518 400 mg b.i.d. | KALETRA™ 400/100 mg b.i.d.
Serious Adverse Events (participants affected / at risk) | 15/174 | 10/174
Other Adverse Events (participants affected / at risk) | 76/174 | 77/174
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | MK0518 400 mg b.i.d. (N=174) | KALETRA™ 400/100 mg b.i.d. (N=174)
Angina pectoris (Cardiac disorders) | 1 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 1
Basedow's disease (Endocrine disorders) | 0 | 1
Ulcerative keratitis (Eye disorders) | 0 | 1
Abdominal pain lower (Gastrointestinal disorders) | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 1
Abdominal abscess (Infections and infestations) | 1 | 0
Appendicitis (Infections and infestations) | 0 | 1
Cellulitis (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 0 | 1
Pneumonia staphylococcal (Infections and infestations) | 1 | 0
Pulmonary tuberculosis (Infections and infestations) | 0 | 1
Pyelonephritis acute (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 1 | 0
Accidental overdose (Injury, poisoning and procedural complications) | 1 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 1 | 0
Foreign body trauma (Injury, poisoning and procedural complications) | 1 | 0
Limb injury (Injury, poisoning and procedural complications) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cerebrospinal fistula (Nervous system disorders) | 1 | 0
Lumbar radiculopathy (Nervous system disorders) | 1 | 0
Acute stress disorder (Psychiatric disorders) | 1 | 0
Bipolar I disorder (Psychiatric disorders) | 1 | 0
Depression (Psychiatric disorders) | 1 | 0
Renal impairment (Renal and urinary disorders) | 1 | 0
Epididymitis (Reproductive system and breast disorders) | 1 | 0
Vasodilatation (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | MK0518 400 mg b.i.d. (N=174) | KALETRA™ 400/100 mg b.i.d. (N=174)
Constipation (Gastrointestinal disorders) | 4 | 3
Diarrhoea (Gastrointestinal disorders) | 9 | 18
Nausea (Gastrointestinal disorders) | 6 | 8
Vomiting (Gastrointestinal disorders) | 2 | 6
Asthenia (General disorders) | 2 | 4
Fatigue (General disorders) | 7 | 7
Influenza like illness (General disorders) | 4 | 3
Bronchitis (Infections and infestations) | 5 | 7
Gastroenteritis (Infections and infestations) | 5 | 2
Influenza (Infections and infestations) | 4 | 6
Nasopharyngitis (Infections and infestations) | 12 | 6
Pharyngitis (Infections and infestations) | 1 | 4
Sinusitis (Infections and infestations) | 5 | 5
Syphilis (Infections and infestations) | 4 | 3
Upper respiratory tract infection (Infections and infestations) | 7 | 5
Alanine aminotransferase increased (Investigations) | 5 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 6 | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 4
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 5
Dizziness (Nervous system disorders) | 6 | 0
Headache (Nervous system disorders) | 10 | 9
Anxiety (Psychiatric disorders) | 5 | 2
Depression (Psychiatric disorders) | 8 | 5
Insomnia (Psychiatric disorders) | 5 | 5
Cough (Respiratory, thoracic and mediastinal disorders) | 5 | 6
Rash (Skin and subcutaneous tissue disorders) | 3 | 5
Hypertension (Vascular disorders) | 4 | 1

LIMITATIONS AND CAVEATS:
The reason for early termination: Study was terminated after the primary efficacy analysis at Week 24 did not demonstrate non-inferiority of MK0518 versus KALETRA™.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Merck agreements may vary with individual investigators, but will not prohibit any investigator from publishing. Merck supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.